CLINICAL TRIAL: NCT03150901
Title: Role of Adiponectine in Pathophysiology Ogf Diabetic Foot
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Marina Shargorodsky, Shargorodsky MARINA, Wolfson Medical Center
Other Study IDs: 0016-15-WOMC
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetic patients: In a prospective study, we will collect wound edge tissue specimens from 75 patients with DF during surgical debridement. From each patient, 1-4 specimens will be obtained per debridement. To evaluate debrided tissue, each specimen will be processed for paraffin embedding and stained with haematoxylin and eosin. Histopathology analysis of multiple specimens acquired from the same wound will be analysed. Full-thickness epidermis biopsies will be followed by biomarker assessment such as:
  1. Expression of insulin-like growth factor 1 receptor (IGF-1R)
  2. Adiponectin
  3. Leptin
  4. Resistin
  5. Osteocalcin
  6. Osteoprotegerin
  7. Insulin, c-peptid
  8. HOMA-IR
  Interventions: Diagnostic Test: no drug

INTERVENTIONS:
Diagnostic Test: no drug — laboratory tests

SUMMARY:
Diabetic patients with a history of diabetic foot are considered to be a high-risk population for increased cardiovascular and all-cause mortality (1,2,3,). Diabetic foot (DF) is responsible for more hospitalizations than any other complication of diabetes and are the leading cause of non-traumatic lower extremity amputations, resulting in nearly 100 000 amputations annually in the US alone (4,5,6). Surgical debridement, as an important component of standard of care of diabetic foot, is intended to remove healing-impaired tissue, decreases bacterial burden, thus to stimulate overall wound closure, while removing as little of healing-competent skin as possible. Furthermore, debrided tissue is often used as a valuable tissue source for research purposes (7,8,9,10). Debrided tissue presents valuable diagnostic and research source to verify pathology, assess prognosis and gain insights into DF molecular pathology, all of which ultimately leads to improved outcomes.

We aimed to validate tissue obtained from surgical debridement of DF for the cellular/molecular tissue analyses and biomarkers, to evaluate the pathophysiology of DF and understanding mechanisms that inhibit healing.

The age range will be 50-70 years, in order to minimize the effects of irreversible vascular wall changes induced progressively by the aging process. All patients will undergo screening procedures that will include full anamnesis, physical examination, basic laboratory blood tests (full chemistry, CBC); urine examination and EKG will be performed at start and at the end of the study. Patients with a significant myocardial, and renal, cerebrovascular or hepatic disease will be excluded from the study.

In a prospective study, we will collect wound edge tissue specimens from 75 patients with DF during surgical debridement. From each patient, 1-4 specimens will be obtained per debridement. To evaluate debrided tissue, each specimen will be processed for paraffin embedding and stained with haematoxylin and eosin. Histopathology analysis of multiple specimens acquired from the same wound will be analysed.

DETAILED DESCRIPTION:
Diabetic patients with a history of diabetic foot are considered to be a high-risk population for increased cardiovascular and all-cause mortality (1,2,3,). Diabetic foot (DF) is responsible for more hospitalizations than any other complication of diabetes and are the leading cause of non-traumatic lower extremity amputations, resulting in nearly 100 000 amputations annually in the US alone (4,5,6). Surgical debridement, as an important component of standard of care of diabetic foot, is intended to remove healing-impaired tissue, decreases bacterial burden, thus to stimulate overall wound closure, while removing as little of healing-competent skin as possible. Furthermore, debrided tissue is often used as a valuable tissue source for research purposes (7,8,9,10). Debrided tissue presents valuable diagnostic and research source to verify pathology, assess prognosis and gain insights into DF molecular pathology, all of which ultimately leads to improved outcomes.

We aimed to validate tissue obtained from surgical debridement of DF for the cellular/molecular tissue analyses and biomarkers, to evaluate the pathophysiology of DF and understanding mechanisms that inhibit healing.

The age range will be 50-70 years, in order to minimize the effects of irreversible vascular wall changes induced progressively by the aging process. All patients will undergo screening procedures that will include full anamnesis, physical examination, basic laboratory blood tests (full chemistry, CBC); urine examination and EKG will be performed at start and at the end of the study. Patients with a significant myocardial, and renal, cerebrovascular or hepatic disease will be excluded from the study.

In a prospective study, we will collect wound edge tissue specimens from 75 patients with DF during surgical debridement. From each patient, 1-4 specimens will be obtained per debridement. To evaluate debrided tissue, each specimen will be processed for paraffin embedding and stained with haematoxylin and eosin. Histopathology analysis of multiple specimens acquired from the same wound will be analysed. Full-thickness epidermis biopsies will be followed by biomarker assessment such as:

1. Expression of insulin-like growth factor 1 receptor (IGF-1R)
2. Adiponectin
3. Leptin
4. Resistin
5. Osteocalcin
6. Osteoprotegerin
7. Insulin, c-peptid
8. HOMA-IR Blood sampling for chemistry and metabolic markers including lipids, fasting glucose, fasting insulin, HbA1C, HOMA-IR , CRP, plasma adiponectin, visfatin, resistin, and plasma leptin will be performed. Additionally, relationship between serum and tissue adipokines level will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized from January 2015 through December 2016 in Wolfson Medical Center due to the diagnosis of diabetic foot

Exclusion Criteria:

* Patients with a history of unstable angina, MI, CVA or major surgery within the six months preceding entrance to the study were excluded.
* Patients with unbalanced endocrine disease were excluded, as were patients with plasma creatinine > 2.5 mg/dl and elevation of liver enzymes to more than twice the upper normal limit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients hospitalized from January 2015 through December 2016 in Wolfson Medical Center due to the diagnosis of diabetic foot
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
dIABETIC FOOT ULCERS INCIDENCE | 1 year

IPD SHARING:
Plan to Share IPD: Undecided